CLINICAL TRIAL: NCT03292107
Title: Study on Management Thrombosis in Greek Cancer Patients (GMaT - Greek Management Thrombosis)
Brief Title: Study on Management Thrombosis in Greek Cancer Patients
Acronym: GMaT
Status: Completed | Type: Observational
Sponsor: Hellenic Society of Medical Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: Management Thrombosis
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study on Management Thrombosis in Greek cancer patients

DETAILED DESCRIPTION:
The approach that Medical Oncologists encounter the prospect of a coagulation event occurrence in cancer patients.

ELIGIBILITY:
Inclusion Criteria

* All patients diagnosed with histologically confirmed solid tumors that are under anticoagulation therapy, during the study timeline.
* Age ≥ 18 years
* Signed informed consent

Exclusion Criteria

* Initiation of anticoagulation therapy before the initiation of the study in 2016
* Age <18 years
* No signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumors under anticoagulation regime, for prophylaxis or treatment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
The clinical practice for patients under anticoagulation regime | 1 YEAR
  Documentation of the clinical practice for patients under anticoagulation regime, for prophylaxis or treatment, in patients with solid tumors, for one year following the protocol initiation date, including high-risk patients as defined in the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Varthalitis, MD, Principal Investigator — Hellenic Society of Medical Oncology
Locations (1):
- Hellenic Society of Medical Oncology, Athens, Greece

REFERENCES:
- [Derived] Christopoulou A, Ardavanis A, Papandreou C, Koumakis G, Papatsimpas G, Papakotoulas P, Tsoukalas N, Andreadis C, Samelis G, Papakostas P, Aravantinos G, Ziras N, Souggleri M, Kalofonos C, Samantas E, Makrantonakis P, Pentheroudakis G, Athanasiadis A, Stergiou H, Bokas A, Grivas A, Tripodaki ES, Varthalitis I, Timotheadou E, Boukovinas I. Prophylaxis of cancer-associated venous thromboembolism with low-molecular-weight heparin-tinzaparin: Real world evidence. Oncol Lett. 2022 Apr;23(4):115. doi: 10.3892/ol.2022.13235. Epub 2022 Feb 9. PMID 35251346